CLINICAL TRIAL: NCT06284434
Title: Liposomal Bupivacaine Use in Alveolar Bone Graft Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kerry O'Rourke (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Sponsor-Investigator, Kerry O'Rourke, Clinical research coordinator, Shriners Hospitals for Children
Organization: Shriners Hospitals for Children (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CHI2311
Record Dates: First submitted 2024-02-21; First posted 2024-02-29 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Cleft Lip and Palate
Keywords: cleft lip; cleft palate; alveolar bone graft; pain management; liposomal bupivacaine
MeSH Terms: conditions — Cleft Lip; Cleft Palate; Agnosia | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: The design of this study is a randomized control trial, double-blinded. Patients who meet criteria and consent will be randomized to receive LB or standard bupivacaine.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Surgeons and patients will be unaware of which cohort the subject will be randomized to be part of. The pharmacist, anesthesiologist, and research coordinator may all be aware of which drug is administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LB Treatment Arm (Experimental): Patients on the treatment arm will receive liposomal bupivacaine mixed with epinephrine (ratio of 1:100,000), which is not considered the standard of care.
  Interventions: Drug: Liposomal Bupivacaine; Drug: Epinephrine
- Bupivacaine Control Arm (Active Comparator): Patients on the control arm will follow the current standard of care, which is traditional bupivacaine mixed with epinephrine (1:100,000).
  Interventions: Drug: Bupivacain; Drug: Epinephrine

INTERVENTIONS:
Drug: Liposomal Bupivacaine — Patients will receive liposomal bupivacaine mixed with epinephrine (ratio of 1:100,000) for pain management after surgery.
  Other Names: EXPAREL
  Arms: LB Treatment Arm
Drug: Bupivacain — Patients will receive standard bupivacaine mixed with epinephrine (ratio of 1:100,000) for pain management after surgery.
  Arms: Bupivacaine Control Arm
Drug: Epinephrine — Patients will receive epinephrine (ratio of 1:100,000) mixed with the appropriate drug assigned to them based on their arm.
  Other Names: Adrenalin

SUMMARY:
The goal of this clinical trial is to learn if a pain medication called liposomal bupivacaine (brand name EXPAREL®) with epinephrine will provide better pain control, increased activity, and reduced use of opioids compared with the standard treatment for patients age 6 years and older with cleft lip and palate who have had an alveolar bone graft surgery. Investigators will look at:

* pain scores at hip and jaw sites
* opioid use in amount and frequency
* scores on activity questionnaires Researchers will compare the results of these items with those of patients who had the standard treatment of bupivacaine with epinephrine.

DETAILED DESCRIPTION:
The study is a randomized, double-blinded trial comparing liposomal bupivacaine (EXPAREL®) with epinephrine (0.25%) local anesthetic with the standard treatment of bupivacaine with epinephrine (0.25%) local anesthetic. The study will enroll patients with cleft lip and palate undergoing an alveolar bone graft (ABG) surgery. Researchers will enroll a maximum of 60 patients from Shriners Children's Chicago over a 2-year period.

After this surgery, patients experience significant pain. Considering both the frequency of reported pain after ABG combined with the current opioid crisis and subsequent recommendations by organizations such as the American Society of Anesthesiologists Task Force on Acute Pain Management and Guidelines from the Society for Pediatric Anesthesia for alternative pain management, the use of liposomal bupivacaine (EXPAREL®) is a potential alternative to reduce post-operative pain in the pediatric ABG population.

Liposomal bupivacaine (LB) is an injectable form of bupivacaine used at the surgical site and that is released over time. Studies have shown that LB better controls pain, especially during the first 24 hours post-surgery. Better pain control has been associated with a reduction in opioid usage and its associated complications.

The study is designed to randomize patients to either the standard of care (bupivacaine with epinephrine) or liposomal bupivacaine with epinephrine to better study pain management within the first five days after ABG surgery in Shriners' cleft lip and palate patients.

The FDA approved EXPAREL® for the adult population in 2011 and for the pediatric population, age 6 years and older in 2021. It is a locally injected single dose analgesia that is released over 72 hours.

The study is considered minimal risk because LB use does not present an increased risk over the standard of care (standard bupivacaine) as it is an alternative form of the same pain medication. Previous studies have shown no additional risk to using the liposomal version of bupivacaine vs standard bupivacaine in ABG surgeries.

Patients will participate up to 5 days following surgery (surgery day is considered day 0) with reported pain, activity scores, and opioid use collected through either paper, electronic, or phone questionnaires. Surgeons and patients will be unaware of which cohort the patient will be randomized to be part of. The pharmacist, anesthesiologist, and research coordinator may all be aware of which drug is administered.

Researchers will obtain informed consent from the participants and/or their legally authorized representatives before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are 6 and older who have a diagnosis of cleft lip and/or palate with a scheduled surgery that involves an alveolar bone graft.

Exclusion Criteria:

* Patients under age 6 are excluded from this study as EXPAREL® is not FDA approved for this group.
* Patients with a history of allergic or adverse reaction to any drug involved in the study (EXPAREL, Epinephrine, or Bupivacaine).
* Patients with a history of cardiovascular disease.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-04-24 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Pain Scores | on Day 1 to Day 5 after surgery
  Pain scores at hip and jaw sites. Pain is rated on a 0 to 10 scale with 0 representing no pain and 10 representing agonizing pain with unbearable distress. A lower score is ideal for improved pain management.
Opioid Use | on Day 1 to Day 5 after surgery
  Opioid use in amount and frequency
PROMIS Pediatric Mobility Questionnaire | on Day 1 to Day 5 after surgery
  The patient will log activity level using the Patient Reported Outcome Measurement Information System (PROMIS) Pediatric Mobility scale. The categorical answers to the questions are the minimum value "not able to do", "with a lot of trouble", "with some trouble", "with a little trouble", and the maximum value "with no trouble." Therefore a higher amount of reported with no trouble categorical answers would represent improved mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Chad A. Purnell, MD, Principal Investigator — Shriners Hospitals for Children
Locations (1):
- Shriners Children's Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chughtai M, Sultan AA, Hudson B, Goodwin RC, Seif J, Khlopas A, Bena J, Jin Y, Gurd DP, Kuivila TE, Ballock RT. Liposomal Bupivacaine Is Both Safe and Effective in Controlling Postoperative Pain After Spinal Surgery in Children: A Controlled Cohort Study. Clin Spine Surg. 2020 Dec;33(10):E533-E538. doi: 10.1097/BSD.0000000000000996. PMID 32324672
- [Background] Crowley JS, McLean P, Gabriel RA, Cronin B, Hsieh S, Englar K, Said E, Lance S, Gosman A. The Association of Liposomal Bupivacaine on Opioid Consumption in the Pediatric Alveolar Cleft Population. J Craniofac Surg. 2020 Jun;31(4):1078-1081. doi: 10.1097/SCS.0000000000006310. PMID 32195834
- [Background] Flowers T, Winters R. Postoperative pain management in pediatric cleft lip and palate repair. Curr Opin Otolaryngol Head Neck Surg. 2021 Aug 1;29(4):294-298. doi: 10.1097/MOO.0000000000000719. PMID 34183559
- [Background] Patel RA, Jablonka EM, Rustad KC, Pridgen BC, Sorice-Virk SS, Borrelli MR, Khosla RK, Lorenz HP, Momeni A, Wan DC. Retrospective cohort-based comparison of intraoperative liposomal bupivacaine versus bupivacaine for donor site iliac crest analgesia during alveolar bone grafting. J Plast Reconstr Aesthet Surg. 2019 Dec;72(12):2056-2063. doi: 10.1016/j.bjps.2019.09.026. Epub 2019 Oct 2. PMID 31648962